CLINICAL TRIAL: NCT02511288
Title: Liquid Biopsies in Patients With Advanced Non-small Cell Lung Cancer
Brief Title: LIquid BIopsies in Patients Presenting Non-small Cell Lung Cancer
Acronym: LIBIL
Status: Recruiting | Type: Observational
Sponsor: Centre Leon Berard (Other)
Responsible Party: Sponsor
Other Study IDs: ET15-076 LIBIL
Record Dates: First submitted 2015-07-16; First posted 2015-07-30 (Estimated); Last update posted 2024-08-21 (Actual); Status verified 2024-08

CONDITIONS: Carcinoma, Non-Small-Cell Lung
Keywords: Hematologic test; Liquid biopsy
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood samples
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- Cohort 1: Patients with advanced NSCLC and no druggable molecular alteration at time of diagnosis
- Cohort 2: Patients with advanced NSCLC harboring targetable molecular alterations at time of diagnosis
- Cohort 3: Patients with advanced NSCLC at time of immunotherapy introduction (1st or 2nd line)

SUMMARY:
The goal of this project is to characterize the genetic profile of patients with advanced stage IIIB/IV non-small cell lung cancer (NSCLC) using liquid biopsies

DETAILED DESCRIPTION:
Lung cancers are the first cause of death by cancer in the world. The majority of these patients are diagnosed at a late stage, non-eligible to a curative treatment. Due to tumoral genomic identification, it has been possible to classify NSCLC in molecular subtypes according to molecular abnormalities detection called "drivers" which can be targeted using an appropriate treatment. This change modifies the standard treatments from the very first line of treatment particularly for patients having an EGFR mutation or an ALK or ROS1 rearrangement, with a significant benefit of progression free survival. The French NCI (INCa) recommends to identify genomic alterations of a genes panel including EGFR, KRAS, BRAF, HER2, ALK and ROS1 as well as mutations in MET exon 14. However, all the patients who benefit from a targeted therapy develop resistance after a mean duration of 10-12 months after starting the treatment. In case of progression, the tumour genetic analysis through new biopsies, enables to identify these mechanisms and then to determine if the patient can benefit or not from a third generation molecule active on these mechanisms, and to have a better understanding of the disease evolution.

The detection of these alterations is routinely performed using tissular biopsies but in 10 to 20% of the cases, it is not possible.

The detection of these molecular abnormalities in the plasma, called " liquid biopsy " is a valuable non-invasive complementary approach for these patients. It is presently used in routine for detecting the EGFR mutations at diagnosis as well as for searching EGFR T790M mutation for resistant patients.

The liquid biopsies enable to detect circulating tumoral DNA.

ELIGIBILITY:
COHORT 1

Inclusion Criteria:

* Patients with histologically confirmed advanced non-small-cell lung carcinoma (stage IIIB/IV) regardless of the mutation status
* Inclusion at the time of diagnostic
* Realization of tumor biopsy at the institution (Centre Léon Bérard) or outside the institution with an available histopathological report
* Age ≥ 18 years
* Covered by a health insurance
* Signed consent

Exclusion Criteria:

- Patients treated before their liquid biopsy

COHORT 2 Inclusion criteria

* Patients with histologically confirmed advanced non-small-cell lung carcinoma (stage IIIB/IV) with one of the following molecular anomalies: Epidermal Growth Factor Receptor (EGFR), B-Raf proto oncogene (BRAF) or Human Epidermal Growth Factor Receptor-2 (HER2) mutations, Anaplatsic Lymphoma Kinase (ALK) or ROS porto-oncogene 1 (ROS1) translocation, Mesenchymal-epithelial transition factor (MET) amplification, RET rearrangement.
* Inclusion at the time of diagnosis
* Realization of tumor biopsy at the institution (Centre Léon Bérard) or outside the institution with an available histopathological report
* Age ≥ 18 years
* Covered by a health insurance
* Signed consent

COHORT 3 Inclusion criteria

* Patients with histologically confirmed advanced non-small-cell lung carcinoma (stage IIIB/IV) whatever the mutational or PD-L1 status.
* Inclusion at the time of immunotherapy treatment initiation (1st or 2nd line)
* Realization of tumor biopsy at the institution (Centre Léon Bérard) or outside the institution with an available histopathological report
* Age ≥ 18 years
* Covered by a health insurance
* Signed consent

Exclusion criteria

- Initiation of immunotherpy before their liquid biopsy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with advanced NSCLC
Sampling Method: Non-Probability Sample
Enrollment: 900 (Estimated)
Dates: Start 2015-07 (Actual); Primary Completion 2026-03 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Identification of the genetic profile in advanced or metastatic NSCLC patients using liquid biopsies (circulating tumoral DNA) | 5 years
  Technique: ddPCR + targeted NGF, whole exome sequencing

SECONDARY OUTCOMES:
Identification of genetic biomarkers (or molecular profiles) having a potential predictive value in the treatments response | 5 years
  Techniques: ddPCR + targeted NGF, whole exome sequencing
Detection of the ALK and ROS1 genes translocations in the circulating DNA | 5 years
  Techniques: ddPCR + targeted NGF, whole exome sequencing
Evaluation of the liquid biopsies role in the tumoral monitoring | 5 years
  Correlation between mutated allelic fractions or expression's modification with the treatment response. Techniques: ddPCR + targeted NGF, whole exome sequencing
Evaluation of genomic and transcriptomic factors detectable in the plasma, associated to the immunotherapy response | 5 years
  Correlation between transcriptomic and genomic factors and response to immunotherapy. Techniques: ddPCR + targeted NGF, whole exome sequencing
Evaluation of the spatial and temporal tumor heterogeneity under targeted therapy treatment | 5 years
  Techniques: ddPCR + targeted NGF, whole exome sequencing
Evaluation of the miRNAs' expression in plasma as an epigenetic factor associated to treatments response | 5 years
  Correlation between miRNAS expression in plasma and treatment's efficacy. Techniques: miRNAs profiling using HTG technology
Circulating tumoral cells isolation and analysis to determine the role of non-genomic and/or phenotypic factors in the treatments response. | 5 years
  Single cell isolation technology
Evaluation of the resistance mechanisms to targeted therapies | 5 years
  Technique: ddPCR + targeted NGF, whole exome sequencing

CONTACTS AND LOCATIONS:
Overall Officials: Pierre Saintigny, MD, PhD, Study Director — pierre.saintigny@lyon.unicancer.fr
Locations (8):
- France (8):
  - Centre Hospitalier Annecy Genevois, Annecy
  - CH Fleyriat, Bourg-en-Bresse
  - Hôpital Louis Pradel, Bron
  - CHU Grenoble Alpes, Grenoble
  - Centre Léon Bérard, Lyon
  - CHRU de Saint-Etienne, Saint-Priest-en-Jarez
  - Institut de Cancérologie Lucien Neuwirth, Saint-Priest-en-Jarez
  - Hôpital Nord Ouest, Villefranche-sur-Saône